CLINICAL TRIAL: NCT06774638
Title: Diagnostic and Prognostic Biomarkers in SARS-CoV-2 Infections
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: MAC-2020
Record Dates: First submitted 2024-12-01; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-10

CONDITIONS: IBD - Inflammatory Bowel Disease; COVID - 19
MeSH Terms: conditions — Inflammatory Bowel Diseases; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Literature data document that SARS-CoV-2 RNA is present not only in the respiratory tract but also in the feces of infected patients, suggesting a potential additional route of transmission: the oro-fecal route. In this context, it becomes essential to have data on the use of serological tests in suspected SARS-CoV-2 patients and the presence of viral RNA in biological samples from affected patients, to quickly and reliably identify infected individuals and provide recommendations on the duration of patient isolation. In particular, such data could support the indication for contact isolation similar to that used for all highly contagious gastrointestinal infections, such as Clostridium difficile, with a longer duration than respiratory isolation. The objective of this study is to verify the presence of diagnostic and prognostic biomarkers in patients with SARS-CoV-2 infection.

DETAILED DESCRIPTION:
- Sample Size Calculation

Given the exploratory nature of the study, no formal sample size calculation was performed. A total of 370 patients is expected to be enrolled.

- Data Analysis (as outlined in the approved protocol)

Data will be analyzed using t-tests (or Mann-Whitney tests, depending on the data type). The correlation between obtained results and clinical outcomes will be tested using Spearman's rank correlation coefficient to identify potential biomarkers.

For microbiota analysis, intra-sample diversity (alpha diversity) will be assessed using Faith's phylogenetic diversity metrics, observed OTUs, and the Shannon index. Inter-sample diversity (beta diversity) will be evaluated using weighted and unweighted UniFrac distances, which will serve as input for principal coordinates analysis (PCoA). PCoA plots, heatmaps, and bar plots will be created using the Made4 and Vegan packages in R. Statistical analysis will be conducted using the Vegan and Stats packages. The separation of data in PCoA will be tested using a permutation test with pseudo-F ratios (Adonis function in Vegan). Fisher's exact test will be used to assess the significance of differences between clusters obtained through hierarchical clustering analysis. The Wilcoxon test (for paired or unpaired data) will be employed to compare alpha and beta diversity, as well as the relative abundance of microbial groups (or functional groups) between subject groups and over time. Discriminatory features (taxa or genes) will be identified using Random Forests (Breiman, 2001). Microbiota sequences from healthy subjects, matched for age, sex, and BMI, will be retrieved from publicly accessible databases for comparative purposes. p-values will be adjusted for multiple comparisons using the Benjamini-Hochberg method. A false discovery rate <0.05 will be considered statistically significant.

Correlations between variables will be assessed using Kendall's correlation test with the cor.test function from the Stats package in R.

For microbiota analysis, intra-sample diversity (alpha diversity) will be assessed using Faith's phylogenetic diversity metrics, observed OTUs, and the Shannon index. Inter-sample diversity (beta diversity) will be evaluated using weighted and unweighted UniFrac distances, which will serve as input for principal coordinates analysis (PCoA). PCoA plots, heatmaps, and bar plots will be created using the Made4 and Vegan packages in R. Statistical analysis will be conducted using the Vegan and Stats packages. The separation of data in PCoA will be tested using a permutation test with pseudo-F ratios (Adonis function in Vegan). Fisher's exact test will be used to assess the significance of differences between clusters obtained through hierarchical clustering analysis. The Wilcoxon test (for paired or unpaired data) will be employed to compare alpha and beta diversity, as well as the relative abundance of microbial groups (or functional groups) between subject groups and over time. Discriminatory features (taxa or genes) will be identified using Random Forests (Breiman, 2001). Microbiota sequences from healthy subjects, matched for age, sex, and BMI, will be retrieved from publicly accessible databases for comparative purposes. p-values will be adjusted for multiple comparisons using the Benjamini-Hochberg method. A false discovery rate <0.05 will be considered statistically significant.

Correlations between variables will be assessed using Kendall's correlation test with the cor.test function from the Stats package in R.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Collection of informed consent to participate in the study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the IBD unit with clinical diagnosis of SARS-CoV-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-04-04 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
The objective of this study is to verify the presence of diagnostic and prognostic biomarkers in patients with SARS-CoV-2 infection. | At baseline, one time, during the hospitalization.
  Evaluate the potential presence and persistence of SARS-CoV-2 RNA in the feces of clinically recovered patients with a negative nasopharyngeal swab.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Gionchetti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy